CLINICAL TRIAL: NCT01214408
Title: Effect of Digene Total on 24 Hrs Ambulatory Gastric ph in Pts Suffering From Acid Peptic Disorder After Single and Repeated Dosing.
Brief Title: Effect of Digene Total (Buffered Pantoprazole) on 24 Hour Gastric Potential Hydrogen (pH) in Patients From Acid Peptic Disorder After Single and Repeated Dosing.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R12-576
Record Dates: First submitted 2010-10-03; First posted 2010-10-05 (Estimated); Last update posted 2012-12-28 (Estimated); Status verified 2012-12

CONDITIONS: Acid Peptic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GRP-A (Experimental)
  Interventions: Drug: Buffered pantoprazole
- GRP-B (Experimental)
  Interventions: Drug: Buffered pantoprazole

INTERVENTIONS:
Drug: Buffered pantoprazole — Buffered pantoprazole 40 mg QD
  Other Names: ABT-897, Buffered Pantoprazole, Digene Total
  Arms: GRP-A
Drug: Buffered pantoprazole — Buffered pantoprazole 40 mg QD
  Other Names: ABT-897, Buffered Pantoprazole, Digene Total
  Arms: GRP-B

SUMMARY:
This prospective, open label, single-center and non-comparative study is designed to generate data on Digene Total's (buffered pantoprazole) rapid and sustained gastric acid inhibition effect in patients suffering from acid peptic disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects (18-65 years) suffering from acid peptic disorder (APD), diagnosed endoscopically (reflux esophagitis, gastritis and peptic ulcer)
2. Must voluntarily sign and date an informed consent form, approved by an Independent Ethics Committee (IEC)/ Institutional Review Board (IRB), prior to any study specific procedures.
3. If female, subject must be either postmenopausal for at least 1 year, surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or practicing at least one of the following methods of birth control:

   1. Total abstinence from sexual intercourse (minimum one completed menstrual cycle)
   2. A vasectomized partner
   3. Hormonal contraceptives (oral, parenteral or transdermal) for at least 3 months prior to study drug administration.
   4. Intrauterine device (IUD)
   5. Double barrier method (condoms, contraceptive sponge, diaphragm or vaginal ring with spermicidal jellies or creams)

Exclusion Criteria:

1. Subjects with concurrent gastrointestinal diseases, gastric surgery, perforation or bleeding
2. Subjects who have a history of use of any antisecretory drug within past 7 days prior study Day 0
3. Subjects with cardiac, neurological, renal or hepatic dysfunction
4. Past history of significant sensitivity or contraindication to study drug
5. Pregnant or breast-feeding female
6. Any condition that, in the opinion of the Investigator, does not justify the subject's inclusion for the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Time taken to achieve a gastric pH of > 4 after a single dose of Digene Total (buffered pantoprazole) | Assessment done on day 1 for group A subjects

SECONDARY OUTCOMES:
Percentage of time gastric pH was > 4 after repeated dosing of Digene Total (buffered pantoprazole) | Assessment done on day 7 for all subjects
24 hour median gastric pH after repeated dosing of Digene Total (buffered pantoprazole) | Assessment done on day 1 for group A subjects

CONTACTS AND LOCATIONS:
Overall Officials: Balagopal Nair, MD, Study Director — Abbott
Locations (1):
- Site Reference ID/Investigator# 42043, Chennai, India

REFERENCES:
- See also: For more information, click on the website link — http://dailymed.nlm.nih.gov/dailymed/about.cfm